CLINICAL TRIAL: NCT03725956
Title: Effects of Endoscopic Sinus Surgery on Sleep Disorder in Patients With Chronic Rhinosinusitis With Polyps
Brief Title: Polysomnographic Findings in Nasal Polyposis
Acronym: POLYSOMNO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018_19; 2018-A01650-55 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-18; First posted 2018-10-31 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Obstructive Sleep Apnea
Keywords: Nasal polyposis; sleep; sinus surgery; polysomnography; quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopic sinus surgery (Experimental): Single group of patients with nasal polyposis eligible for endoscopic sinus surgery
  Interventions: Procedure: Endoscopic sinus surgery

INTERVENTIONS:
Procedure: Endoscopic sinus surgery — Surgical procedure under general anaesthesia:
  Consists of the removal of bone boundaries between sinus cavities (ethmoidectomy) with nasal polyps resection in order to retrieve nasal patency and sinus drainage Polysomnographic assessment as routinely applied in clinical practice

SUMMARY:
Nasal polyposis (NP) is a chronic inflammatory disease of the nasal and sinus mucosa leading to protrusion of edematous polyps in the nasal cavity. Prevalence of NP among the chronic rhinosinusitis patients is 25-30 %. NP leads to significant limitations in physical, emotional and social aspects of life of the affected patients. Sleep disorder is frequently reported by those patients with impaired nasal breathing. Till now few studies have objectively assessed the impact of NP on sleep quality. the objectives are to figure out sleep disturbances in NP and to analyze the outcomes of sinus surgery on sleep recovering.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic sinus surgery for recalcitrant nasal polyposis (failure of a 4-month corticosteroid medical treatment) Social insured patient
* Patient willing to comply with all procedures of the study and its duration
* Patient giving consent

Exclusion Criteria:

* Patients with previous nasal surgery for nasal polyposis
* Patients with previous continuous positive airway pressure therapy for obstructive sleep apnea
* Non-coverage by the social security scheme
* Patient unable to receive informed information
* Refusal to sign the consent
* Person deprived of the liberty
* Person benefiting from a system of legal protection (guardianship…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Slow-wave sleep duration | 1 month before surgery and 3 months postoperatively
  Slow-wave sleep duration is measured one month before surgery and 3 months after surgery

SECONDARY OUTCOMES:
change in total sleep duration | At 1 month before surgery and at 3 months postoperatively
Change in the number of brief wakefulness | At 1 month before surgery and at 3 months postoperatively
change in Apnea-hypopnea index | At 1 month before surgery and at 3 months postoperatively
  This index measures the number of apnea and hypopnea during the total sleep duration.
Change in time with oxygen desaturation below 90% | At 1 month before surgery and at 3 months postoperatively
change in Epworth sleepiness scale scores | At 1 month before surgery and at 3 months postoperatively
  The Epworth sleepiness scale score is a questionnaire based of 8 questions assessing daytime sleepiness. Each question is graded from 0 to 3. A total score ranging from 0 to 24 is established:
  1 to 6 points: Normal sleep 7 to 8 points: Average sleepiness 9 to 24 points: Abnormal (possibly pathologic) sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Mortuaire, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France